CLINICAL TRIAL: NCT02456818
Title: A Hospital-based Cohort Study in German Hematological / Oncological Wards to Assess the Effect of Contact Isolation on Nosocomial Colonization With ESBL-producing Escherichia Coli (CONTAIN Study)
Brief Title: Assessing the Effect of Contact Isolation on Nosocomial Colonization With ESBL-EC in German Hematology/Oncology Wards
Acronym: CONTAIN
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Cologne (Other)
Collaborators: University Hospital Tuebingen (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital, Aachen (Other)
Responsible Party: Principal Investigator, Maria J.G.T. Vehreschild, PD Dr.med, University of Cologne
Other Study IDs: CONTAIN
Record Dates: First submitted 2015-02-24; First posted 2015-05-29 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Oncology [See Also, Affected System]; Hematological Disease; Infection Due to ESBL Escherichia Coli
Keywords: Colonization; Multi-resistant gram negative bacteria; Infection control measures; Hand hygiene program; Contact precautions; Immunocompromised host
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Rectal swabs or stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Centers using contact isolation: * Isolation triggered by the detection of ESBL-EC at hospital admission in surveillance screening or during the hospitalization by weekly screening or clinical cultures
  * Contact isolation terminated, after at least two negative consecutive fecal screening cultures
  * Contact isolation resumed, if subsequent ESBL-EC positive cultures are identified for the same patient including readmissions
  Contact isolation must include:
  * Patient placement in single rooms
  * Cohorting only possible, when no single rooms available and corresponding ESBL-EC strains are phenotypically identical
  * Staff and visitors wearing gloves and gowns as contact precautions when entering the room, patient when leaving the room
- Centers using no contact isolation: * not regularly isolating for ESBL-EC
  * ESBL-EC colonized or infected patients with urinary or fecal incontinence or diarrhea (>3 loose bowel movements/day) isolated in single rooms with above described contact precautions

SUMMARY:
This study aims to evaluate the impact of contact isolation on the rate of hospital-acquired transmissions of ESBL-producing Escherichia coli (ESBL-EC) and the rate of colonization and infection. On the basis of this study, it will be possible to re-evaluate the need for contact isolation for patients colonized or infected with ESBL-EC.

DETAILED DESCRIPTION:
The study aims to evaluate the impact of contact isolation on the rate of hospital-acquired transmissions of ESBL-producing Escherichia coli and the rate of colonization and infection.

Hematological and oncological wards in hospitals with a non-outbreak setting for ESBL-EC and adhering to at least the following standard of care are eligible for study participation:

* Fecal screening for the presence of ESBL-EC of all patients within 72 hours of each admission by use of a rectal swab or stool sample
* Follow-up fecal screening once a week and within 72 hours of discharge
* Implementation of clinical standards aimed at ESBL-EC decolonization is not allowed on wards participating in this study, including in the context of clinical studies.

Sites will be grouped according to their approach regarding contact isolation (see group description).

As a control for external factors a hand hygiene program, including training and adherence assessments, will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Wards adhering to at least the following standard of care are eligible for study participation:
* Fecal screening for the presence of ESBL-EC of all patients within 72 hours of each admission by use of a rectal swab or stool sample
* Follow-up fecal screening once a week and within 72 hours of discharge

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All admitted patients on participating hematological and oncological wards in hospitals with a non-outbreak setting for ESBL-EC.
Sampling Method: Non-Probability Sample
Enrollment: 2264 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of hospital-acquired ESBL-EC colonization or infection | up to 12 month

SECONDARY OUTCOMES:
Incidence of patient-to-patient transmission of ESBL-EC defined by the isolation of two or more ESBL-EC strains from two or more different patients with overlapping hospitalization periods in the same ward, related to each other on the basis of molecular | up to 12 month
Incidence of ESBL-EC intestinal colonization among all patients (colonization is defined as the isolation of ESBL-EC in material from fecal screening) | up to 12 month
Incidence of ESBL-EC bloodstream infections among all patients (ESBL-EC bloodstream infection is defined by the isolation of ESBL-EC from blood cultures) | up to 12 month
Incidence of ESBL-EC bloodstream infections among previously colonized patients - Readmission fraction associated with infection with ESBL-EC | up to 12 month
Incidence of ESBL-Klebsiella pneumonia (ESBL-KP) colonized patients among all patients (colonization is defined as the isolation of ESBL-KP in material from fecal screening) | up to 12 month
  In theory, the ability to produce ESBL can be transferred between species by plasmids. However, in clinical practice, this seems to be an extremely rare event. Nevertheless, it should be assessed to detect any potential risks to patients at sites not isolating for ESBL-EC.
Incidence of ESBL-KP bloodstream infections among all patients (ESBL-EC bloodstream infection is defined by the isolation of ESBL-KP from blood cultures) | up to 12 month
  In theory, the ability to produce ESBL can be transferred between species by plasmids. However, in clinical practice, this seems to be an extremely rare event. Nevertheless, it should be assessed to detect any potential risks to patients at sites not isolating for ESBL-EC.
Incidence of ESBL-KP bloodstream infections among previously colonized patients | up to 12 month
  In theory, the ability to produce ESBL can be transferred between species by plasmids. However, in clinical practice, this seems to be an extremely rare event. Nevertheless, it should be assessed to detect any potential risks to patients at sites not isolating for ESBL-EC.

CONTACTS AND LOCATIONS:
Overall Officials: Maria JG Vehreschild, PD Dr., Principal Investigator — university clinic of cologne; Oliver A Cornely, Prof Dr., Principal Investigator — university clinic of cologne; Jörg J Vehreschild, PD Dr., Principal Investigator — university clinic of cologne; Harald Seifert, Prof. Dr., Principal Investigator — university clinic of cologne